CLINICAL TRIAL: NCT06546410
Title: A Retrospective Multisite Analysis of Routinely Collected Outpatient EEGs for Identifying Seizure Susceptibility in Paediatric Epilepsy Using Computational Biomarkers.
Brief Title: OASIS: RetrOspective Analysis on EEGs for Identifying Seizure Susceptibility in paediatrIcs Using biomarkerS
Acronym: OASIS
Status: Not yet recruiting | Type: Observational
Sponsor: Neuronostics Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: NNBioEP005
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Epilepsy; Epilepsy in Children
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Epilepsy
  Interventions: Device: BioEP
- Non-epilepsy
  Interventions: Device: BioEP

INTERVENTIONS:
Device: BioEP — All patient's EEG will have the BioEP score conducted on it

SUMMARY:
The goal of this retrospective study is to validate a set of computational biomarkers (BioEP) for seizure susceptibility on retrospective routinely collected non-contributory EEGs in paediatric participants with epilepsy. The main objectives are:

Primary:

To validate a set of computational biomarkers (BioEP) for seizure susceptibility on retrospective routinely collected non-contributory EEGs in paediatric participants with epilepsy.

Secondary:

To examine whether the use of BioEP could support a more efficient patient pathway to diagnosis (thus adding economic value), by reducing time to final diagnosis and/or the number of clinical appointments needed

ELIGIBILITY:
Inclusion Criteria:

* ≥2-<18 years age.
* Patients who have had a confirmed epilepsy diagnosis for ≥1+ year.
* Non contributary first EEG: including routine EEG, sleep EEG (natural, melatonin induced, sleep deprived), 24-hour ambulatory EEG.
* Patients who have been diagnosed with a self-limited and or focal epilepsy [*] who have had a first non-contributary (no IEDS present, negative) outpatient EEG.
* Patients who have been diagnosed with idiopathic generalised epilepsy [†] who have had a first non-contributary (no IEDS present, negative) routine EEG.
* Neurodiverse patients with epilepsy can be included in the study [‡]
* Patients with epilepsy and co-morbidities can be included in the study (anxiety, mood disorders etc)
* Controls should be EEGs taken from patients who have been referred for a paroxysmal disorder, received an EEG as part of their diagnostic work up and subsequently received an alternate diagnosis. Epilepsy should have been excluded from their differential diagnosis and the alternate diagnosis should have remained stable for ≥1+ year.

Exclusion Criteria:

* Developmental and/or epileptic encephalopathies [§]
* Patients with global development delay of unknown origin.
* Patients with profound and multiple intellectual disabilities
* Participants with a known hepatic/renal encephalopathy.
* Patient diagnosed with possible NEAD and epilepsy (dual diagnosis).
* Participants taking part in another Clinical Trial of an Investigational Medicinal Product (CTIMP) (qualitative/observational studies are acceptable).
* Patients with any breaches of skull (plates, burr holes, shrapnel).

Ages: 2 Years to 16 Years | Sex: All
Age Groups: Child
Study Population: Paediatric population with a diagnosis of epilepsy.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
To validate a set of computational biomarkers (BioEP) for seizure susceptibility on retrospective routinely collected non-contributory EEGs in paediatric participants with epilepsy. | 1 year
  We shall demonstrate biomarkers from those with epilepsy are distinct from controls by measuring levels of balanced accuracy (sensitivity, specificity, positive predictive ratio, negative predictive ratio, diagnostic odds ratio, and area under operator curve characteristics curve)

SECONDARY OUTCOMES:
To examine whether the use of BioEP could support a more efficient patient pathway to diagnosis (thus adding economic value), by reducing time to final diagnosis and/or the number of clinical appointments needed | 1 year
  Reduction in time and cost to patients with the use of BioEP

CONTACTS AND LOCATIONS:
Overall Officials: Milaana Mainstone, Study Director — Neuronostics Ltd

IPD SHARING:
Plan to Share IPD: Undecided